CLINICAL TRIAL: NCT03984760
Title: A Multicenter, Randomized, Open-Label, Active-Controlled, Parallel Study to Assess the Efficacy and Safety of Ferric Citrate Capsules for the Treatment of Hyperphosphatemia in Patients With Chronic Kidney Disease Undergoing Hemodialysis
Brief Title: Ferric Citrate for the Treatment of Hyperphosphatemia in Patients With Chronic Kidney Disease Undergoing Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Panion & BF Biotech Inc. (Industry)
Collaborators: Shandong Weigao Panion Pharmaceutical Co. Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WG-PBB00302
Record Dates: First submitted 2019-06-05; First posted 2019-06-13 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Hyperphosphatemia; End Stage Renal Disease; ESRD
Keywords: Kidney Diseases; Kidney Failure, Chronic; Hyperphosphatemia; Renal Insufficiency, Chronic; Renal Insufficiency; Phosphorus Metabolism Disorder
MeSH Terms: conditions — Hyperphosphatemia; Kidney Failure, Chronic; Kidney Diseases; Renal Insufficiency, Chronic; Renal Insufficiency; Phosphorus Metabolism Disorders | interventions — ferric citrate; Sevelamer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ferric Citrate Capsule (Experimental): Ferric Citrate Capsule, product specification: 500 mg/cap, manufactured by Panion & BF Biotech Inc.
  Interventions: Drug: Ferric Citrate
- Sevelamer Carbonate Tablet (Active Comparator): Sevelamer carbonate tablet group, product specification: 800 mg/tablet, manufactured by Genzyme Ireland Limited
  Interventions: Drug: Sevelamer Carbonate

INTERVENTIONS:
Drug: Ferric Citrate — Take the capsules with meals or immediately after meals.
  Arms: Ferric Citrate Capsule
Drug: Sevelamer Carbonate — Take the tablets with meals.
  Arms: Sevelamer Carbonate Tablet

SUMMARY:
To evaluate the efficacy and safety of ferric citrate capsules for the treatment of hyperphosphatemia in patients with chronic kidney disease undergoing hemodialysis

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label, active-controlled, parallel, phase III study which aims to assess the efficacy and safety of ferric citrate capsules for the treatment of hyperphosphatemia in patients with chronic kidney disease undergoing hemodialysis. This study is consisting of a Screening/Washout period (14 days) and a Treatment/Observation period (12 weeks). During the Treatment period, the subjects will be randomly assigned to the ferric citrate capsule group (study group) or sevelamer carbonate tablet group (control group) in the ratio of 1:1.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to give written informed consent.;
2. Between the age of 18 and 75 years (including the boundary value);
3. Patients who maintain the hemodialysis schedule as 3 times a week and the dialysis schedule should remain unchanged during the study period;
4. At Screening, patients who have received phosphate binder for at least 4 weeks and have a serum phosphorus level between 2.5 and 8.0 mg/dL (0.81 to 2.58 mmol/L) (excluding the boundary value) after treatment;
5. Patients with a serum phosphorus level between 5.5 and 10.0 mg/dL (1.78 to 3.23 mmol/L) (excluding the boundary value) after washout.

Exclusion Criteria:

1. Patients with severe gastrointestinal diseases (such as acute peptic ulcer, chronic ulcerative colitis, regional enteritis, ileus) or patients with dysphagia;
2. Patients with a history of gastrectomy or enterectomy (excluding endoscopic excision or caecectomy) or patients who had undergone gastrointestinal surgery within 3 months prior to Screening;
3. Patients with severe constipation (times of bowel movement≤ 1 time/week), chronic diarrhea (times of bowel movement≥ 4 times/day), severe gastrointestinal motility disorder;
4. Patients with hemochromatosis or patients receiving treatment for iron overload, or patients with a serum ferritin level >800 ng/mL or TSAT >50% at Screening;
5. Patients with a serum calcium level (corrected) <8.0 mg/dL (2.0 mmol/L) or >11.0 mg/dL (2.75 mmol/L) after washout;
6. Patients with intact-PTH>800pg/mL at Screening, or patients undergone parathyroid surgery within 6 months prior to Screening or requiring parathyroid surgery;
7. Patients who received blood transfusions for treating anemia within 3 months prior to Screening;
8. Patients who require phosphorus-binding agents containing aluminum, magnesium, calcium and lanthanum in addition to the study drug or patients who require an antacid with a phosphorus binding effect during the study period;
9. Patients who require citrate preparation as an anticoagulant during hemodialysis treatment during the study period;
10. Patients with impaired liver function (hepatic dysfunction or serum total bilirubin, aspartate aminotransferase or alanine aminotransferase ≥ 2 times the upper limit of normal) or patients with cirrhosis;
11. Patients with cerebrovascular disease (cerebral infarction, cerebral hemorrhage, etc.) or cardiovascular disease (congestive heart failure of Class III or severer in NYHA classification, acute myocardial infarction, unstable angina, etc.) requiring hospitalization within 6 months prior to Screening;
12. Patients who are known to be intolerant to sevelamer carbonate tablet;
13. Patients with a history of allergies to iron preparations or those who are intolerant to iron preparations;
14. Patients who are scheduled to have a kidney transplant during the study period;
15. Patients with a current or past history of malignancy within 5 years prior to Screening;
16. Women who are pregnant or lactating, or patients who are unable to take effective contraception from screening to 6 months after discontinuation (including male subjects and their female spouses);
17. Patients who had participated in other clinical studies and other received investigational drug product within 1 month or 5 half-lives of the drug product (whichever is longer) prior to Screening;
18. Patients who are not suitable for participating in the trial according to the investigator's judgment;
19. Patients who are unwilling or unable to follow the protocol process.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
The change in serum phosphorus levels | 12 Weeks
  The change in serum phosphorus levels at the end of treatment (Visit 10 or ET) as compared to baseline (before the first dose).

SECONDARY OUTCOMES:
Serum phosphorus levels | 12 Weeks
  Serum phosphorus levels at the end of treatment;
The proportion of subjects whose serum phosphorus levels reached the target range. | 12 Weeks
  The proportion of subjects whose serum phosphorus levels reached the target range (3.5 to 5.5 mg/dL, 1.13 to 1.78 mmol/L) at the end of the treatment;
The response rate of serum phosphorus | 12 Weeks
  The response rate of serum phosphorus at the end of treatment (defined as reduction of the serum phosphorus level exceeds 25% as compared to baseline);
The change in serum calcium (corrected) levels | 12 Weeks
  The change in serum calcium (corrected) levels at the end of treatment as compared to baseline;
The change in the [Ca] × [P] product relative | 12 Weeks
  The change in the [Ca] × [P] product relative at the end of treatment as compared to baseline;
The change in the level of intact-PTH levels | 12 Weeks
  The change in the level of intact-PTH levels at the end of treatment as compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangmei Chen, Principal Investigator — The General Hospital of the People's Liberation Army (PLAGH)
Locations (24):
- China (24):
  - Baotou Central Hospital, Baotou
  - The General Hospital of the People's Liberation Army (PLAGH), Beijing
  - The Second Hospital of Jilin University, Changchun
  - Daping Hospital, Chongqing
  - The First Affiliated Hospital of Dalian Medical University, Dalian
  - The Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The First Affiliated Hospital/School Of Clinical Medicine of Guangdong Pharmaceutical University, Guangzhou
  - Jilin Guowen Hospital, Jilin
  - Jiujiang University Affiliated Hospital, Jiujiang
  - Meihekou Central Hospital, Meihekou
  - Jiangxi Provincial People's Hospital, Nanchang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - BenQ Medical Center, Nanjing
  - JiangSu Province Hospital (The First Affiliated Hospital of Nanjing Medical University), Nanjing
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Changhai Hospital, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - Tonghua Central Hospital, Tonghua
  - Fifth Hospital in Wuhan, Wuhan
  - Renmin Hospital of Wuhan University, Wuhan
  - Zhongnan Hospital of Wuhan University, Wuhan
  - Henan Provincial People's Hospital, Zhengzhou
  - Affiliated Hospital of Zunyi Medical University, Zunyi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086